CLINICAL TRIAL: NCT00022776
Title: Randomized Clinical Trial of Treatment for Spinal Stenosis
Brief Title: Surgical Versus Nonsurgical Treatment for Spinal Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01 AR45633; R01AR045622 (NIH)
Record Dates: First submitted 2001-08-13; First posted 2001-08-15 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Spinal Stenosis
Keywords: Human therapy evaluation; Orthopedics; Physical therapy; Nonsurgical treatment; Surgical decompression; Surgery; Lumbar; Spine disorder; Spinal stenosis; Gender difference; Medical rehabilitation
MeSH Terms: conditions — Spinal Stenosis; Spinal Diseases | interventions — Decompression, Surgical; Laminectomy; Foraminotomy; Physical Therapy Modalities; Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will undergo surgery for spinal stenosis. Participants in this group will undergo surgical decompression as described by Rothman and Simeone.
  Interventions: Procedure: Surgical decompression
- 2 (Experimental): Participants will undergo physical therapy for spinal stenosis. These participants will undergo a physical therapy program emphasizing lumbar flexion exercises, general conditioning exercises, and patient education for six weeks, with a frequency of 1-2 visits per week. Each patient will receive instruction in a home exercise program.
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Surgical decompression — Simple decompression not requiring fusion.
  Other Names: Laminectomy; Foraminotomy
  Arms: 1
Procedure: Physical therapy — 2 physical therapy sessions per week for 6 weeks Followed by home program.
  Other Names: Exercises; Aerobics; Strengthening
  Arms: 2

SUMMARY:
Lumbar spinal stenosis (a narrowing of spaces in the backbone that results in pressure on the spinal cord and/or nerve roots) is a condition that occurs frequently, particularly in the elderly. This condition can lead to significant pain and limit a person's ability to function. Moreover, doctors disagree about the best way to treat people with lumbar spinal stenosis.

In this study we will compare surgical treatment of lumbar spinal stenosis with nonsurgical treatment using physical therapy. The results of this study should help clarify which treatment strategies are the most effective for patients with lumbar spinal stenosis.

DETAILED DESCRIPTION:
Lumbar spinal stenosis is a frequently encountered condition, particularly in the elderly, which can lead to significant pain and functional limitations. The prevalence of this condition is growing as the population continues to age. Substantial controversy exists regarding the management of lumbar spinal stenosis. Surgery has traditionally been the treatment of choice, although physicians typically recommend a trial of nonsurgical care prior to surgery. The most effective means of nonsurgical treatment has not been identified, although a "standard" regimen has been developed.

There is presently no evidence in the literature regarding the relative effectiveness of surgical versus nonsurgical treatment of lumbar spinal stenosis, or the efficacy of the standard nonsurgical treatment approach. This randomized clinical trial will compare surgical decompression versus nonsurgical treatment (i.e., physical therapy) of lumbar spinal stenosis. The results of this study should help clarify which treatment strategies are the most effective for patients with lumbar spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Imaging evidence of stenosis
* Unable to walk more than 1/4 of a mile
* No prior surgery for stenosis
* Consents to surgery
* Speaks English

Exclusion Criteria:

* Presence of dementia or organic brain syndrome
* Coronary artery disease, recent myocardial infarction, pulmonary or vascular disease
* Spondylolisthesis (> 5 mm slippage)
* Severe osteoporosis
* Metastatic cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2000-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study 36-item Short Form Health Survey | Measured at Month 24

SECONDARY OUTCOMES:
Beck Depression Inventory | Measured at Month 24
Oswestry Low Back Pain Disability Scale | Measured at Month 24
MODEMS questionnaires | Measured at Month 24
Physical impairments and function, including lower leg strength, reflexes, walking tolerance on a treadmill, and two-stage treadmill test | Measured at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Delitto, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Delitto A, Piva SR, Moore CG, Fritz JM, Wisniewski SR, Josbeno DA, Fye M, Welch WC. Surgery versus nonsurgical treatment of lumbar spinal stenosis: a randomized trial. Ann Intern Med. 2015 Apr 7;162(7):465-73. doi: 10.7326/M14-1420. PMID 25844995